CLINICAL TRIAL: NCT00077051
Title: Translational Phase I Trial of Escalating Doses of 5-Chloro-2'-Deoxycytidine (CldC) With a Fixed Dose of Tetrahydrouridine Combined With a Fixed Dose of Cisplatin Concomitant With Definitive Radiation in Patients With Advanced Squamous Cell Carcinoma of the Oral Cavity and Oropharynx
Brief Title: Cytochlor and Tetrahydrouridine as Radiosensitizers and Cisplatin Combined With Radiation Therapy in Treating Patients With Advanced Squamous Cell Carcinoma of the Oral Cavity (Mouth) or Oropharynx (Throat)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20020154; SCCC-2002033; NCI-6301
Record Dates: First submitted 2004-02-10; First posted 2004-02-11 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Tetrahydrouridine; Radiotherapy

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: cisplatin; Drug: cytochlor; Drug: tetrahydrouridine; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin
Drug: cytochlor
Drug: tetrahydrouridine
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Radiosensitizing drugs, such as cytochlor and tetrahydrouridine, may make tumor cells more sensitive to radiation therapy. Drugs used in chemotherapy, such as cisplatin work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Combining radiosensitizers with chemotherapy and radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of cytochlor when given together with tetrahydrouridine, cisplatin and radiation therapy in treating patients with advanced squamous cell carcinoma of the oral cavity (mouth) or oropharynx (throat).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose range of cytochlor to be used in phase II trials, based on safety, toxicity, and tissue selectivity, in patients with advanced squamous cell carcinoma of the oral cavity or oropharynx.
* Determine the safety and toxicity profile of cytochlor, tetrahydrouridine, and concurrent radiotherapy followed by radiotherapy alone in these patients.
* Determine the percentage of cancer cells vs normal cells that incorporate cytochlor in the DNA of patients treated with this regimen.
* Determine the percentage replacement of thymine by 5-chlorouracil in tumors vs normal tissue of patients treated with this regimen.

Secondary

* Determine the tissue selectivity of this regimen in these patients.
* Determine the level of cytochlor and its metabolites within the serum and urine of these patients during combination treatment and before radiotherapy alone is initiated.
* Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is an open-label, dose-escalation study of cytochlor.

Patients receive tetrahydrouridine IV over 5 minutes followed by cytochlor IV for 3 days on week 1 and 5 days a week on weeks 2-4 and cisplatin IV over 30-60 minutes once in weeks 2 and 5. Patients also undergo radiotherapy 5 days a week during weeks 2-7. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of cytochlor until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 1 of 3 or 3 of 6 patients experience dose-limiting toxicity.

Patients are followed at 1 month, monthly for 3 months, every 3 months for up to 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 3-18 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell carcinoma of the oral cavity or oropharynx

  * Stage III disease not eligible for surgery
  * Stage IV disease allowed if patient is not eligible for chemotherapy or refused chemotherapy
  * No distant metastasis
* Previously untreated disease
* No osteoradionecrosis in patients with tumors involving the maxilla
* Tumor tissue/normal adjacent tissue (T/N) ratio for dC kinase and dCMP deaminase greater than 2.5

PATIENT CHARACTERISTICS:

Age

* Over 21

Performance status

* Karnofsky 80-100% OR
* ECOG 0-1

Life expectancy

* More than 6 months

Hematopoietic

* Absolute neutrophil count greater than 1,500/mm^3
* WBC at least 3,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic

* AST/ALT less than 2.5 times upper limit of normal
* Bilirubin normal

Renal

* Creatinine normal OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No impending carotid rupture

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study treatment
* HIV negative
* No other concurrent uncontrolled illness
* No active or ongoing infection
* No alcohol dependence
* No psychiatric illness or social situation that would preclude study compliance
* No other malignancy within the past 3 years except low-risk, non-melanomatous skin cancer, carcinoma in situ (e.g., breast, cervix, or bladder), or stage T1-2, low-to-moderate grade prostate cancer (Gleason score no greater than 7)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent hormonal therapy except contraceptives or replacement steroids

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Other

* No prior therapy for head and neck cancer
* No other concurrent experimental medications
* No other concurrent anticancer therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2004-04; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis E. Raez, MD, FACP, Study Chair — University of Miami Sylvester Comprehensive Cancer Center; May Abdel-Wahab, MD, PhD, Principal Investigator — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida, United States